CLINICAL TRIAL: NCT00781989
Title: Qualification of Ultrasonography as a Biomarker of Prognosis and Response to Treatment in Early Rheumatoid Arthritis
Brief Title: Ultrasonography as a Biomarker in Early Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: CRO1089; Sponsers number: TAYP2013; Funder's number: G0601962
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis
Keywords: early rheumatoid arthritis; biomarkers; ultrasound
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood / serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis patients: Patients with seropositive Rheumatoid Arthritis with symptom onset of less than three years

SUMMARY:
This is a prospective, observational study designed to look at ultrasound images of the joint at baseline and over time, and investigate whether there is a correlation between ultrasound images and progression of disease. The researchers wish also to see if ultrasound can be used as a tool to predict progression of Rheumatoid Arthritis in patients with early disease who have not taken biologics therapy. In addition, the researchers wish to investigate whether peripheral blood "biomarkers"can be identified that predict the progression of erosive disease in early rheumatoid arthritis, with the intention of testing the most promising biomarkers in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 18 years or greater.
2. The subject has a diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology (ACR) with onset of symptomatology of less than 3 years.
3. The patient is seropositive for rheumatoid factor (IgM RF measured by agglutination assay) and / or anti-cyclic citrullinated peptides (measured by ELISA).
4. The subject has provided signed and dated written informed consent prior to admission to the study
5. The subject is able to understand and comply with protocol requirements, instructions and restrictions.

Exclusion Criteria:

1. Past or present disease, which as judged by the investigator, may affect both the subject's participation in the study or outcome of the study. These diseases include but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease.
2. Current or prior use of biologic drugs ( anti- tumour necrosis factor alpha drugs or rituximab)
3. As a result of the medical interview, physical examination or screening investigations, the physician responsible considers the subject unfit for the study.
4. The subject's RA does not have a clearly recordable time of onset (within a 6 month period) as determined by either the notes or from the history taken from the patient by the physician responsible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital Rheumatology outpatient departments
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Correlation between Power Doppler Ultrasound (PDUS)score at baseline and progression of erosions at one year, as assessed by xray and high frequency ultrasound. | one year

SECONDARY OUTCOMES:
Correlation between average Power Doppler Ultrasound (PDUS) score (at 0,6 and 12 months) and progression of erosions at one year,as assessed by xray and high frequency ultrasound. | one year
Correlation between CRP level at baseline and progression of erosions at one year,as assessed by xray and high frequency ultrasound. | one year

CONTACTS AND LOCATIONS:
Overall Officials: P C Taylor, MA, PhD, Principal Investigator — Imperial College London
Locations (1):
- Kennedy Institute Clinical Trials Unit, 4 West, Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sreerangaiah D, Grayer M, Fisher BA, Ho M, Abraham S, Taylor PC. Quantitative power Doppler ultrasound measures of peripheral joint synovitis in poor prognosis early rheumatoid arthritis predict radiographic progression. Rheumatology (Oxford). 2016 Jan;55(1):89-93. doi: 10.1093/rheumatology/kev305. Epub 2015 Aug 27. PMID 26316580